CLINICAL TRIAL: NCT03329456
Title: Minimum Effective Volume (MEV95%) of Ropivacaine 7.5 mg/ml to Block the Posterior and Lateral Cords of the Infraclavicular Brachial Plexus
Brief Title: MEV to Block the Posterior and Lateral Cords of the Infraclavicular Brachial Plexus
Acronym: LSIB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Musso
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2017-10

CONDITIONS: Shoulder Disease; Anesthesia
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ropivacaine (Other): Single arm intervention
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Minimum effective volume

SUMMARY:
The investigators have recently shown that LSIB in combination with a suprascapular and a cervical plexus block is a very good alternative for arthroscopic shoulder surgery. However, the investigators believe the total volume of local anesthetic for LSIB may be reduced. For shoulder surgery there is no need to block the medial cord and the investigators therefore hypothesize a significantly lower MEV95% by applying a selective lateral and posterior cord block

DETAILED DESCRIPTION:
The MEV for a successful block in 50% of the participants will be determined by using the staircase up-and-down method introduced by Dixon and Massey. Logistic regression and probit transformation will be applied to estimate the MEV for a successful block in 95% of the participants.

ELIGIBILITY:
Inclusion Criteria:

* . Inclusion criteria are American Society of Anesthesiologists (ASA) physical status I-III, age between 18 and 70 years and body mass index (BMI) between 20 and 35 kg/m2.

Exclusion Criteria:

* Exclusion criteria are pregnancy, patients with contraindications to regional anesthesia, allergy to LAs, patients taking opioids regularly due to chronic pain, use of anticoagulation drugs other than acetylsalicylic acid or dipyridamole, atrioventricular block, diabetes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Minimum effective volume (95%) | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lars M Ytrebø, M.D Ph.D, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Musso D, Flohr-Madsen S, Meknas K, Wilsgaard T, Ytrebo LM, Klaastad O. A novel combination of peripheral nerve blocks for arthroscopic shoulder surgery. Acta Anaesthesiol Scand. 2017 Oct;61(9):1192-1202. doi: 10.1111/aas.12948. Epub 2017 Aug 4. PMID 28776638
- [Derived] Musso D, Klaastad O, Wilsgaard T, Ytrebo LM. Brachial plexus block of the posterior and the lateral cord using ropivacaine 7.5 mg/mL. Acta Anaesthesiol Scand. 2019 Mar;63(3):389-395. doi: 10.1111/aas.13277. Epub 2018 Oct 18. PMID 30338518